CLINICAL TRIAL: NCT00677079
Title: A Phase 2, Single Arm Study of BSI-201 in Patients With BRCA-1 or BRCA-2 Associated Advanced Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Single Arm Study of BSI-201 in Patients With BRCA-1 or BRCA-2 Associated Advanced Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD11489; 20080105 (Other: BiPar)
Expanded Access: NCT01130259 (No longer available)
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Primary Peritoneal Cancer; Advanced Epithelial Ovarian Cancer
Keywords: BRCA-1 or BRCA-2 associated advanced epithelial ovarian, fallopian tube, or primary peritoneal cancer; BRCA-1; BRCA-2
MeSH Terms: conditions — Fanconi Anemia, Complementation Group D1 | interventions — iniparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iniparib (Experimental): Iniparib, twice weekly on Days 1 and 4 of each week during 8-week cycles
  Interventions: Drug: Iniparib

INTERVENTIONS:
Drug: Iniparib — Body weight adjusted dose
  1 hour intravenous infusion
  Other Names: BSI-201; SAR240550

SUMMARY:
The goal of this study was to determine the efficacy of iniparib (BSI-201/SAR240550) in patients with breast cancer gene-associated (BRCA) ovarian cancer.

Up to 35 patients were to be treated using a Simon 2-stage optimal design, i.e. twelve were to be treated in a first stage, then if 2/12 patients responded to treatment as defined by Response Evaluation Criteria in Solid Tumor (RECIST), 23 additional patients were be treated in the second stage.

DETAILED DESCRIPTION:
Participants were treated for at least one 8-week cycle, with additional cycles as long as they had stable or responding disease (per RECIST criteria) and wished to remain on study.

Participants had a final follow-up visit within 4 weeks following the last dose of iniparib, after which time they were contacted by study staff every 3 months for the first year and every 6 months thereafter to assess disease status and survival.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 or older;
* Histologically or cytologically confirmed advanced epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer (stage III or IV);
* At least one previous regimen with platinum/taxane combination therapy and no curative options as determined by their physician (no limit on the number of prior therapies);
* Confirmed BRCA1 or BRCA2 status;
* One or more measurable lesions, at least 10mm in longest diameter by spiral computed tomography (CT) scan or 20mm in longest diameter when measured with conventional techniques (palpation, plain x-ray, CT or magnetic resonance imaging (MRI));
* Karnofsky performance status ≥70%;
* Estimated life expectancy of at least 16 weeks.

Exclusion Criteria:

* Normal clinical laboratory values;
* Any anti-cancer therapy within 21 days prior to study start;
* Any other malignancy within 3 years of study start, except adequately treated carcinoma in situ of the cervix, ductal carcinoma in situ (DCIS) of the breast, or basal or squamous cell skin cancer;
* Active viral infection including HIV/AIDS, Hepatitis B or Hepatitis C infection;
* Active central nervous system or brain metastases;
* History of seizures or current treatment with anti-epileptic medication;
* Persistent grade 2 or greater toxicities from prior therapy, excluding alopecia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Best overall response | until treatment discontinuation (assessment at the at the end of each 8-week cycle)
  Best overall response was defined as the best evaluation observed through the entire treatment period based on Response Evaluation Criteria in Solid Tumor (RECIST) criteria.
Objective response rate | until treatment discontinuation (assessment at the at the end of each 8-week cycle)
  Objective response rate was defined as the percentage of participants with confirmed partial response or complete response according to RECIST criteria.

SECONDARY OUTCOMES:
Clinical benefit rate | until treatment discontinuation (assessment at the at the end of each 8-week cycle)
  Clinical benefit rate was defined as the percentage of participants with complete response, partial response or stable disease according to RECIST criteria.
Progression-Free Survival | until death or study end
  Progression-free survival was defined as the time interval from study entry until disease progression or death due to any cause, whichever came first.
  In the absence disease progression or death, progression-free survival was censored at the last date the participant was known to be alive.
Overall Survival | until death or study end
  Overall Survival was defined as the time interval from study entry until death due to any cause.
  In the absence of confirmation of death, progression-free survival was censored at the last date the participant was known to be alive.
Cancer antigen 125 response (participants with elevated CA125) | until treatment discontinuation (assessment at the at the end of each 8-week cycle)
  Objective response rate was defined as the percentage of participants with confirmed partial response or complete response according to CA125 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- New York, New York, United States

REFERENCES:
- [Derived] Bell-McGuinn KM, Konner JA, Tew WP, Hensley ML, Iasonos A, Charpentier E, Mironov S, Sabbatini P, Aghajanian C. A Phase 2, Single Arm Study of Iniparib in Patients With BRCA1 or BRCA2 Associated Advanced Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer. Int J Gynecol Cancer. 2016 Feb;26(2):255-60. doi: 10.1097/IGC.0000000000000591. PMID 26745694